CLINICAL TRIAL: NCT02212392
Title: COMPARING THE OUTCOME IN PATIENTS OF ACUTE PANCREATITIS, WITH AND WITHOUT PROPHYLACTIC ANTIBIOTICS.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Benazir Bhutto Hospital, Rawalpindi (Other Government)
Responsible Party: Principal Investigator, Dr.Fazal hussain Shah, Resident General surgery, Benazir Bhutto Hospital, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ap3
Record Dates: First submitted 2014-08-05; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Meropenem

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): This arm was not given any prophylactic antibiotics. Patients were managed in the surgical ward by post graduate residents under the supervision of consultants
- Antibiotics (Experimental): this arm was given IV antibiotics, prophylactically, right from the day of admission. They were given intravenous broad spectrum (MEROPENEM) twice daily at 12 hours interval for 7-10 days
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Meropenem — inj. MEROPENEM IV 1 gram twice daily at 12 hours interval for 7-10 days
  Arms: Antibiotics

SUMMARY:
The use of prophylactic antibiotics is beneficial in reducing the extrapancreatic infections and shorter hospital stay in patients of acute pancreatitis as compared to controls.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is an acute inflammatory condition of the pancreas that may extend to local and distant extra pancreatic tissues. AP is broadly classified as mild or severe. Most cases of AP are mild with excellent recovery. However 15% to 20% are severe. Bacterial infections play a vital in the course of the disease. Patients with AP are prone to develop extrapancreatic infections like urinary, respiratory and systemic infections. These infections may result in a prolonged hospitalization, systemic inflammatory response syndrome (SIRS), multi-organ system failure and death. The most common causes are gallstones and alcohol intake. AP is managed by intravenous fluids, analgesia and nothing by mouth. However treatment of severe pancreatitis can be challenging, particularly if multiple organ systems are involved or if there are local complications. In severe acute pancreatitis, as pancreatic enzymes and inflammatory mediators damage the blood vessels and leads to extravasation of fluid in to third space. This fluid extravasation leads to local pancreatic necrosis and end-organ failure. Assessment of severity begins in the emergency room or on admission. Signs of SIRS (high or low core body temperature, tachycardia, tachypnea, low or high peripheral white blood cell count) or organ failure (e.g. elevated serum creatinine) are present on admission in 21% of patients with acute pancreatitis. CT should be considered about 3 days after the onset of symptoms rather than immediately upon admission. Eighty per cent of cases of AP are interstitial and mild; the remaining 20% are necrotizing and severe.

The role of prophylactic antibiotics in acute pancreatitis is controversial .A study published in American Journal of Gastroenterology shows results favouring use of antibiotics in acute pancreatitis. This study shows significant reduction in the length of hospitalization in patients who were given prophylactic antibiotics.

Other Internationally conducted studies suggests that there is no or insignificant role of antibiotics for mild acute pancreatitis and role of prophylactic antibiotics in sever acute pancreatitis for better clinical outcome is controversial to say the least.

Rationale of this study was to emphasize that prophylactic antibiotics in patients with acute pancreatitis can improve patient's out come in terms of shorter hospital stay, and reduced number of extrapancreatic infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 70 years of age with diagnosis of acute pancreatitis both mild and sever necrotizing pancreatitis.
* Patients who present within 48 hours of onset of symptoms.

Exclusion Criteria:

* Patients who present after 48 hours of onset of symptoms.
* Patients already taking antibiotics.
* Patients who are immune compromised
* Patients with debilitating illness i.e. tuberculosis, chronic liver disease.
* Patients with trauma, and multiple visceral injuries
* Patients with diagnosed malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Extrapancreatic infections | 14 days
  it includes infections other than pancreas.It includes the bronchopulmonary infections and the urinary tract infection. Cultures of blood ,urine and sputum was performed in patients who develop fever ˃380C and high peripheral white blood count (leucocytosis ≥10,000/mm3) on blood complete picture. The cultures isolated the organism responsible for the infection.
Duration of hospital stay | average 2 weeks.
  It will be measured in terms of mean number of days (i.e. from the day of admission in surgical ward to the day of discharge.)

CONTACTS AND LOCATIONS:
Overall Officials: Fazal H Shah, MBBS, FCPS I, Principal Investigator — Benazir Bhutto Hospital, Rawalpindi; Sohail Rashid, MBBS, FCPS, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Bilal Altaf, MBBS, FCPS I, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Muhammad Hanif, MBBS, FCPS, Study Chair — Benazir Bhutto Hospital, Rawalpindi
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

REFERENCES:
- [Background] Garcia-Barrasa A, Borobia FG, Pallares R, Jorba R, Poves I, Busquets J, Fabregat J. A double-blind, placebo-controlled trial of ciprofloxacin prophylaxis in patients with acute necrotizing pancreatitis. J Gastrointest Surg. 2009 Apr;13(4):768-74. doi: 10.1007/s11605-008-0773-7. Epub 2008 Dec 11. PMID 19082671
- [Background] Bhopal FG, Azhar F, Mahmood S, Iqbal M. Acute pancreatitis; management, morbidity and mortality experience in a surgical unit. Professional Med J 2011;18: 001-007
- [Background] Cullimore J, Cotter L, Gonzalez A. Antibiotics in acute necrotising pancreatitis. Lancet. 2008 Mar 29;371(9618):1072; author reply 1072. doi: 10.1016/S0140-6736(08)60483-3. No abstract available. PMID 18374839
- [Background] Stevens T, Parsi MA, Walsh RM. Acute pancreatitis: problems in adherence to guidelines. Cleve Clin J Med. 2009 Dec;76(12):697-704. doi: 10.3949/ccjm.76a.09060. PMID 19952294
- [Background] Manes G, Uomo I, Menchise A, Rabitti PG, Ferrara EC, Uomo G. Timing of antibiotic prophylaxis in acute pancreatitis: a controlled randomized study with meropenem. Am J Gastroenterol. 2006 Jun;101(6):1348-53. doi: 10.1111/j.1572-0241.2006.00567.x. PMID 16771960
- [Background] Xue P, Deng LH, Zhang ZD, Yang XN, Wan MH, Song B, Xia Q. Effect of antibiotic prophylaxis on acute necrotizing pancreatitis: results of a randomized controlled trial. J Gastroenterol Hepatol. 2009 May;24(5):736-42. doi: 10.1111/j.1440-1746.2008.05758.x. Epub 2009 Feb 12. PMID 19220676